CLINICAL TRIAL: NCT04572347
Title: National Nurses Health Cohort Study (NNHS): a Web-based Ambispective Cohort Study in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NNHC_1
Record Dates: First submitted 2020-09-30; First posted 2020-10-01 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-09

CONDITIONS: Nurse Health
Keywords: psychophysical health; career development; stress; metabolic indexes
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nurses working in PUTH: Participants will be recruited from Peking University Third Hospital through cluster sampling. Female registered nurses, licensed practical nurses and/or midwives with informed consent are included in this study. The exclusion criteria are student nurses and training nurses.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — It is an observational study, and no intervention will be provided.

SUMMARY:
The purpose of the current study was to build an ambispective cohort study of female nurses, based on existing physical examination and nurse work schedule data and a web-based questionnaire system, focusing on the effects of occupational, environmental, and lifestyle risk factors on the health of Chinese women.

ELIGIBILITY:
Inclusion Criteria:

* Female registered nurses, licensed practical nurses and/or midwives with informed consent are included in this study

Exclusion Criteria:

* student nurses
* training nurses

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from Peking University Third Hospital through cluster sampling.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
psychophysical health related events | From 2010 to 2022
  psychophysical health related events will be collected by web-based questionnaire and hospital information system.
mental health | From 2020 to 2022
  National Aeronautics and Space Administration Task Load Index was used to evaluate the mental workload every year.

SECONDARY OUTCOMES:
sleep quality | From 2020 to 2022
  Pittsburgh sleep quality index was used to evaluate the sleep quality every year.
social support | From 2020 to 2022
  Self developed perceived social support scale was used to evaluate the level of social support every year.

CONTACTS AND LOCATIONS:
Overall Officials: Baohua Li, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yu M, Chen H, Pei M, Zhan S, Li B. Bidirectional Association of Tinnitus and Psychological Distress Among Nurses at One-year Follow-up: A Propensity Score-matched Cohort Study From China. Asian Nurs Res (Korean Soc Nurs Sci). 2025 Dec;19(5):418-425. doi: 10.1016/j.anr.2025.06.003. Epub 2025 Sep 2. PMID 40907657
- [Derived] Che Y, Tang R, Zhang H, Yang M, Geng R, Zhuo L, Wang P, Hu X, Zhou Y, Wang P, Zhan S, Li B. Development of a prediction model for predicting the prevalence of nonalcoholic fatty liver disease in Chinese nurses: the first-year follow data of a web-based ambispective cohort study. BMC Gastroenterol. 2024 Feb 14;24(1):72. doi: 10.1186/s12876-024-03121-1. PMID 38355421
- [Derived] Zhang H, Wang J, Zhang S, Tong S, Hu J, Che Y, Zhuo L, Wang P, Geng R, Zhou Y, Wang P, Zhan S, Li B. Relationship between night shift and sleep problems, risk of metabolic abnormalities of nurses: a 2 years follow-up retrospective analysis in the National Nurse Health Study (NNHS). Int Arch Occup Environ Health. 2023 Dec;96(10):1361-1371. doi: 10.1007/s00420-023-02014-2. Epub 2023 Oct 24. PMID 37874403
- [Derived] Zhuo L, Zhang H, Geng R, Wang P, Zeng L, Che Y, Wang P, Li P, Huang T, Li B, Zhan S. Protocol for the National Nurse Health Study (NNHS): a web-based ambispective cohort study. BMJ Open. 2021 Aug 19;11(8):e049958. doi: 10.1136/bmjopen-2021-049958. PMID 34413106